CLINICAL TRIAL: NCT03041519
Title: Multi-center, Randomized, Controlled, Prospective Trial to Compare the Feasibility, Safety, and Efficacy of Zero-fluoroscopic Ablation Versus Conventional Fluoroscopic Ablation for the Treatment of Ventricular Arrhythmias.
Brief Title: Zero-fluoroscopic Ablation Versus Conventional Fluoroscopic Ablation for the Treatment of Ventricular Arrhythmias
Acronym: ZFOVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Xinyang Central Hospital (Other); Ningbo No. 1 Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yan Wang, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHXXG-ZF-VT-20161220
Record Dates: First submitted 2017-01-29; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Ventricular Arrythmia; Ventricular Premature Complexes; Ventricular Tachycardia
Keywords: Fluoroscopy; Ablation; Three dimensional; Ventricular arrhythmias; Radiation
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zero-fluoroscopy ablation (Experimental): Zero-fluoroscopy ablation will be performed under the guidance of Ensite NavX for mapping and ablation and fluoroscopy will not be used during the procedure.
  Interventions: Procedure: Zero-fluoroscopy ablation
- Conventional fluoroscopy ablation (Active Comparator): Conventional fluoroscopy ablation will be performed under fluoroscopic guidance plus Ensite NavX for mapping and ablation during the procedure.
  Interventions: Procedure: Conventional fluoroscopy ablation

INTERVENTIONS:
Procedure: Zero-fluoroscopy ablation — Catheter ablation will be performed under the guidance of Ensite NavX and without fluoroscopy.
  Arms: Zero-fluoroscopy ablation
Procedure: Conventional fluoroscopy ablation — Catheter ablation will be performed under the guidance of fluoroscopy pllus Ensite NavX.
  Arms: Conventional fluoroscopy ablation

SUMMARY:
This study is intended to compare the feasibility, safety and efficacy of a zero-fluoroscopy approach using Ensite NavX as the only imaging modality with conventional fluoroscopic approach for the catheter ablation of idiopathic ventricular arrhythmias; conventional fluoroscopic approach use fluoroscopy plus Ensite NavX or plus Carto as the imaging modality.

DETAILED DESCRIPTION:
Catheter ablation is a well-established treatment to treat patients with a wide range of heart rhythm disturbances. Fluoroscopy is a imaging modality routinely used for the ablation of arrhythmias.Due to the rising concern regarding the harmful effects of radiation exposure to both the patients and operation staffs; three-dimensional mapping systems, including CARTO and Ensite NavX, have been developed and implemented in electrophysiological procedure for the navigation of catheters inside the heart chambers. Ensite NavX system can be used for zero-fluoroscopy approach for catheter ablation of arrhythmias. This study is intended to compare the feasibility, safety and efficacy of a zero-fluoroscopy approach using Ensite NavX as the only imaging modality with conventional fluoroscopic approach for the catheter ablation of idiopathic ventricular arrhythmias; conventional fluoroscopic approach use fluoroscopy plus Ensite NavX or plus Carto as the imaging modality.

ELIGIBILITY:
Inclusion Criteria:

* Ventricular Tachycardia
* Ventricular Premature Complexes

Exclusion Criteria:

* Organic ventricular tachycardia or ventricular premature complexes
* Drug-induced ventricular tachycardia or ventricular premature complexes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Procedural success rates | 3 months

SECONDARY OUTCOMES:
Total procedure time | during procedure
Fluoroscopy time | during procedure
Complications | 1 year
Immediate success rate | 10~30minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade JG, Rivard L, Macle L. The past, the present, and the future of cardiac arrhythmia ablation. Can J Cardiol. 2014 Dec;30(12 Suppl):S431-41. doi: 10.1016/j.cjca.2014.07.731. Epub 2014 Jul 24. PMID 25432138
- [Background] Anselmino M, Sillano D, Casolati D, Ferraris F, Scaglione M, Gaita F. A new electrophysiology era: zero fluoroscopy. J Cardiovasc Med (Hagerstown). 2013 Mar;14(3):221-7. doi: 10.2459/JCM.0b013e3283536555. PMID 22526222
- [Background] Kozluk E, Gawrysiak M, Piatkowska A, Lodzinski P, Kiliszek M, Malkowska S, Zaczek R, Piatkowski R, Opolski G, Kozlowski D. Radiofrequency ablation without the use of fluoroscopy - in what kind of patients is it feasible? Arch Med Sci. 2013 Oct 31;9(5):821-5. doi: 10.5114/aoms.2013.38676. Epub 2013 Nov 5. PMID 24273563